CLINICAL TRIAL: NCT06532630
Title: An Exploratory Clinical Study Evaluating the Safety and Efficacy of Anti-CD19-CAR-T Cell Therapy in Subjects With Relapsed/Refractory B Cell Malignancies
Brief Title: Anti-CD19-CAR-T Cells in Subjects With Relapsed/Refractory B Cell Malignancies
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai First Song Biotechnology Co., LTD (Industry)
Collaborators: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD19-CN-A5
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-07

CONDITIONS: B-Cell Malignancy
MeSH Terms: interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anti-CD19-CAR-T cell therapy (Experimental): Investigational product: anti-CD19-CAR-T cells.
  Route of administration: Intravenous injection.
  Lymphodepleting chemotherapy regimen: A combination of fludarabine and cyclophosphamide will be administered prior to anti-CD19-CAR-T cells infusion.
  Interventions: Genetic: Anti-CD19-CAR-T cells; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Genetic: Anti-CD19-CAR-T cells — Each subject will be infused with single dose of anti-CD19-CAR-T cells.
  A classic "3+3" dose escalation will be employed.
Drug: Fludarabine — Fludarabine will be given at a dose of 25 mg/m2/day intravenously (IV) for 3 days prior to anti-CD19-CAR-T cells infusion.
Drug: Cyclophosphamide — Cyclophosphamide will be given at a dose of 250 mg/m2/day intravenously (IV) for 3 days prior to anti-CD19-CAR-T cells infusion.

SUMMARY:
This is a single-center, single-arm, open-label, exploratory study to determine the safety, tolerability, feasibility, and preliminary anti-tumor activity of anti-CD19-CAR-T cells in subjects with relapsed/refractory (r/r) B-cell malignancies.

This study plans to enroll patients with relapsed/refractory CD19-positive B-cell malignancies, who will receive a single infusion of anti-CD19-CAR-T cells after screening, PBMC collection, and lymphodepleting chemotherapy.

DETAILED DESCRIPTION:
This study will enroll subjects with CD19-positive relapsed/refractory B-cell malignancies. The effectiveness assessments for anti-CD19-CAR-T cell therapy is evaluated according to international criteria including the 2018 Lugano Classification. Toxicity is evaluated based on the Common Terminology Criteria for Adverse Events (CTCAE, version 5.0) from the National Cancer Institute. The safety of anti-CD19-CAR-T cell therapy will be evaluated through laboratory tests, 12-lead EKGs, and vital signs monitoring. Additionally, blood samples from subjects will be collected to study cellular metabolism and explore the effects of cell therapy on ferritin, C-reactive protein, and related cytokines.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria for inclusion in the study:

1. Patient able to provide written informed consent; parent or guardian of minor patient able to provide written informed consent; ability and willingness to adhere to the study visit schedule and all protocol requirements.
2. 14 - 70 years old.
3. Relapsed/refractory disease after standard treatment (including allogeneic/autologous hematopoietic stem cell transplantation) and not eligible for other treatment options such as a second hematopoietic stem cell transplant.

   A. Relapsed/refractory B-cell acute lymphoblastic leukemia (ALL) is defined as one of the following:
   * Primary refractory disease.
   * Relapsed within 12 months after first remission.
   * Relapsed or refractory after two or more lines of systemic therapy.
   * Relapsed or refractory post allogeneic SCT. i. more than 100 days from the transplantation at the time of enrollment. ii. not receiving immunosuppressive drugs for 4 weeks prior to enrollment (≤5 mg prednisone or equivalent is allowed).

   B. Ph+ B-cell ALL are eligible if they are intolerant or ineligible for tyrosine kinase inhibitor (TKI) therapy or have relapse/refractory disease after at least two different TKI treatments.

   C. Relapsed/refractory B-cell non-Hodgkin lymphoma (NHL) is defined as one of the following:
   1. No response to first-line therapy (primary refractory disease, excluding subjects intolerant to first-line therapy):

      * PD is the best response after first-line therapy.
      * Best response after at least 4 cycles of first-line therapy (e.g., 4 cycles of R-CHOP) is stable disease (SD), with rapid progression in 6 months.
   2. No response to second or subsequent lines of therapy:

      * PD is the best response to last regimen.
      * Best response after at least 2 cycles of the last-line therapy is SD, with rapid progression in 6 months.
   3. Refractory post-autologous stem cell transplant (ASCT):

      * Disease progression or relapse within 12 months (relapse must be biopsy-proven).
      * If salvage therapy is given post-ASCT, the subject must have had no response to or relapsed after the last line of therapy
      * Relapsed or refractory after two or more lines of systemic therapy.
4. Bone marrow with ≥ 5% lymphoblasts by morphologic assessment at screening
5. Relapsed/refractory NHL as one of the following subtypes:

   A. DLBCL-NOS B. Primary mediastinal large B-cell lymphoma (PMBCL) C. Transformed follicular lymphoma (TFL) following prior chemotherapy for follicular lymphoma and subsequent transformation to DLBCL with refractory disease.

   D. Mantle cell lymphoma E. High-grade B-cell lymphoma F. CLL/SLL
6. ECOG performance status ≤2.
7. Life expectancy ≥ 12 weeks.
8. Adequate venous access (for apheresis) and no other contraindications for blood cell separation.
9. Subjects must meet the following laboratory criteria at screening, and they should not have received any growth factors within the 7 days prior to the hematologic assessment:

   A. Absolute neutrophil count ≥1.0×10^9/L. For subjects with ALL, specific criteria will be determined by the investigator.

   B. Hemoglobin ≥60 g/L (without RBC transfusion within 14 days). C. Platelets ≥50×10^9/L. For subjects with ALL, specific criteria will be determined by the investigator.

   D. Absolute lymphocyte count (ALC) ≥0.5×10^9/L. If the total lymphocyte count is insufficient with a high proportion of T cells, the investigator may discuss with the sponsor.

   E. Total bilirubin <1.5×ULN; if liver involved, total bilirubin <3.0×ULN is allowed.

   F. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN; if liver involved, ALT/AST ≤5×ULN is allowed.

   G. Creatinine <1.5×ULN and estimated creatinine clearance ≥60 mL/min.
10. Cardiac ejection fraction (EF) ≥45% with no clinically significant findings on electrocardiogram.
11. Baseline oxygen saturation >92% on room air.
12. Women of childbearing potential must have a negative serum or urine pregnancy test (women who have undergone surgical sterilization or have been postmenopausal for at least 2 years are not considered of childbearing potential).

Exclusion Criteria:

If patients meet any of the following conditions, they cannot participate in this trial:

1. Central nervous system (CNS) involvement in ALL and clinically significant neurological changes (CNS-2 and CNS-3):

   1. CNS-3, defined as detectable tumor cells in cerebrospinal fluid (CSF) with ≥ 5 white blood cells (WBCs) /mm3.
   2. CNS-2, defined as detectable tumor cells in CSF with <5 WBCs /mm3. Note: Subjects with CNS-1 (no detectable tumor cells in CSF) or CNS-2 without evidence of clinically significant neurological changes are eligible for this study.
2. CNS lymphoma confirmed by MRI; active CNS DLBL unless CNS involvement has been effectively treated (i.e., asymptomatic) and a local treatment interval of > 4 weeks prior to enrollment.
3. Active CNS diseases such as epilepsy, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disorders, or any autoimmune diseases involving the central nervous system.
4. Any malignancies other than CD19+ malignancies.
5. Clinically significant heart disease or arrhythmias not controlled by medication.
6. Ongoing or suspected fungal, bacterial, viral, or other infections that are uncontrolled or require intravenous antibiotic therapy; simple urinary tract infections and simple bacterial pharyngitis are allowed.
7. Hepatitis B (positive for hepatitis B surface antigen and hepatitis B DNA >1000 copies/mL) and hepatitis C (positive for hepatitis C antibodies); syphilis, human immunodeficiency virus (HIV) infection.
8. Presence of any indwelling or drainage catheter (e.g., percutaneous nephrostomy, indwelling Foley catheter, biliary drainage catheter, pleural/peritoneal/pericardial drainage catheter); the use of dedicated central venous access devices such as Port-A-Cath® or Hickman® catheters is allowed.
9. Prior use of the following:

   1. CD19-targeted therapy.
   2. Chlorambucil or bendamustine within 3 months before enrollment, or PEG-asparaginase within 3 weeks before enrollment.
   3. live vaccines within 4 weeks before enrollment.
   4. Donor lymphocyte infusions (DLI) within 4 weeks before enrollment.
   5. Medications for graft-versus-host disease (GVHD) treatment within 4 weeks before enrollment, such as calcineurin inhibitors, methotrexate, mycophenolate, rapamycin, or siltuximab, or use of immunosuppressive antibodies (anti-CD20, anti-tumor necrosis factor, anti-interleukin 6, or anti-interleukin 6 receptor) within 4 weeks before enrollment.
   6. Immunostimulatory or immunosuppressive therapy within 4 weeks before enrollment, including interferon-α, interferon-β, IL-2, lenalidomide, efalizumab, alemtuzumab, tocilizumab, cyclosporine, or thalidomide.
   7. Anti-PD-1/anti-PD-L1 therapy within 4 weeks before enrollment.
   8. Systemic cytotoxic chemotherapy within 14 days before enrollment, including daily or weekly low-dose maintenance chemotherapy (e.g., cyclophosphamide, ifosfamide, bendamustine, chlorambucil, melphalan, or vincristine).
   9. Long-acting growth factors (e.g., pegfilgrastim) within 14 days before apheresis or short-acting growth factors within 5 days before apheresis or mobilization agents (e.g., filgrastim/pegfilgrastim, plerixafor) within 5 days before apheresis.
   10. Radiation therapy within 14 days before enrollment.
   11. Pharmacological doses of corticosteroids (>5 mg/day prednisone or equivalent) or other immunosuppressive drugs within 7 days before enrollment.
   12. Venetoclax (BCL-2 inhibitor) within 4 days before apheresis.
   13. Short-acting targeted therapy (e.g., tyrosine kinase inhibitors) within 72 hours before apheresis.
   14. Idelalisib (oral PI3Kδ inhibitor) within 2 days before apheresis.
   15. Lenalidomide within 1 day before enrollment.
10. ≥ Grade 2 graft-versus-host disease (GVHD) per the CIBMTR grading system or requiring systemic corticosteroid treatment exceeding physiological doses.
11. A history of autoimmune diseases in the past 2 years, such as Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus, leading to end-organ damage or requiring systemic immunosuppression or disease-modifying agents.
12. A history of heart attack, cardiac catheterization or stent implantation, unstable angina, or other clinically significant heart diseases within 12 months before enrollment.
13. A history of genetic syndrome with bone marrow failure, such as Fanconi anemia, Kostmann syndrome, Schwachman-Diamond syndrome, etc.
14. Symptomatic deep vein thrombosis or pulmonary embolism requiring systemic anticoagulation within 6 months before enrollment. Subjects need to be on prophylactic anticoagulation.
15. A history of or currently having other malignant tumors (excluding skin basal cell carcinoma, breast/cervical carcinoma in situ, and other malignant tumors that have not been treated in the past five years but are effectively controlled).
16. Use of other investigational medicinal products within 30 days before screening.
17. Pregnant, planning to become pregnant, or breastfeeding in reproductive-aged women. Women who have undergone surgical sterilization or have been postmenopausal for at least 2 years are not considered to be of reproductive potential.
18. Male and female subjects unwilling to practice contraception from the time of agreeing to treatment until 12 months after completion of conditioning chemotherapy or CAR-T infusion.
19. Any past medical history that may interfere with the safety of the study treatment or the evaluation of efficacy.
20. Based on the investigator's judgment, subjects are unlikely to complete all the study visits or procedures required by the protocol.
21. Previous use of any CAR-T cell product or other gene-modified T cell therapy.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-08-24 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerance | 28 days after anti-CD19-CAR-T cells infusion
  Incidence of dose-limiting toxicity (DLT)
Manufacturing feasibility | 1 year
  Percentage of subjects for whom the required dose of anti-CD19-CAR-T cells can be successfully manufactured.

CONTACTS AND LOCATIONS:
Overall Officials: Ge, Study Chair — Thr First Affiliated Hospital of Anhui Medical University; Jian Ge, MD, Principal Investigator — The First Affiliated Hospital of Anhui Medical University
Locations (1):
- The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No